CLINICAL TRIAL: NCT04089917
Title: An Observational Study of the Q Aspiration Catheter Used During Neurointervention for Acute Large Vessel Ischemic Stroke in Spain.
Brief Title: A Study of the Use of the Q Aspiration Catheter to Remove Clot in Stroke Patients
Acronym: TAPAS
Status: Completed | Type: Observational
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 101347
Record Dates: First submitted 2019-08-21; First posted 2019-09-13 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Ischemic
Keywords: Mechanical thrombectomy; Acute ischemic stroke; neurovascular intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Q Aspiration Catheter: mechanical thrombectomy for acute ischemic stroke
  Interventions: Device: Q Aspiration Catheter

INTERVENTIONS:
Device: Q Aspiration Catheter — The Q Aspiration Catheter is indicated for use in the removal of fresh, soft emboli and thrombi in the neurovascular system.

SUMMARY:
The purpose of this study is to collect real-world safety and performance data on the MIVI Neuroscience, Inc. Q Aspiration Catheter for use in the removal of fresh, soft emboli and thrombi in the neurovascular system during acute ischemic stroke.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and performance of the MIVI Neuroscience, Inc. CE Marked Q Aspiration Catheter for use in the removal of fresh, soft emboli and thrombi in the neurovascular system during acute ischemic stroke. The study is an observational study collecting Q Aspiration Catheter use that will enroll a maximum of 50 subjects at a maximum of 5 sites in Spain. Subjects data will be collected through hospitalization with a 3 months post-procedure study visit. This study is designed for observational data to be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years;
* Diagnosis of acute ischemic stroke with mechanical thrombectomy procedure < 8 hours from onset of symptoms/ last known well;
* Large Vessel Occlusion on CT or MRI in the anterior cerebral vasculature up to A1, M1, or M2 or the posterior cerebral vasculature;
* ASPECTS 6 - 10 or volume of diffusion restriction < 50 mL;
* Use of the Q Aspiration Catheter as the first line treatment according to the IFU;
* Signed informed consent by patient or legally authorized representative.

Exclusion Criteria:

* Occlusions in multiple vascular territories, extracranial occlusion or tandem occlusion;
* Evidence of dissection in the carotid or target artery for treatment;
* Evidence of recent/fresh haemorrhage on presentation;
* Unwilling to agree to a 3-month follow up visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population is patients diagnosed with large vessel occlusion acute ischemic stroke within 8 hours of stroke onset treated with mechanical aspiration thrombectomy with the Q Aspiration Catheter as first line therapy.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Espinosa de Rueda Ruiz, MD, Principal Investigator — Neurorradiologia Intervencionista, HCUVA, Murcia
Locations (4):
- Spain (4):
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Centro Hospitalario Universitario Donostia, San Sebastián
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Espinosa de Rueda M, Ballenilla Marco F, Garmendia Lopetegui E, Pumar JM, Zamarro J, Garcia-Villalba B, Diaz-Perez J, Mosqueira A, Luttich A, Larrea JA, Parrilla G. Thrombectomy aspiration post-market study in acute stroke with the Q aspiration catheter: the TAPAS study. J Neurointerv Surg. 2023 Jul;15(7):674-678. doi: 10.1136/neurintsurg-2022-018649. Epub 2022 May 31. PMID 35641183
- See also: Thrombectomy aspiration post-market study in acute stroke with the Q aspiration catheter: the TAPAS study — https://jnis.bmj.com/content/early/2022/05/31/neurintsurg-2022-018649

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Q Aspiration Catheter
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 45

OUTCOME MEASURES:

1. Primary Outcome: Successful Revascularization Rate
Description: Defined as final modified Thrombolysis In Cerebral Infarction scale (mTICI 2b-3) flow in the target vessel
Time Frame: intra-procedural
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Participants | 42

2. Primary Outcome: Symptomatic Intracranial Haemorrhage Rate
Description: Defined as the symptomatic intracranial haemorrhage as detected by CT/MRI with an NIHSS change of >/= 4 points
Time Frame: 24 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Participants | 1

3. Secondary Outcome: Successful Revascularization Rate Using the Q Aspiration Catheter as the Only Thrombectomy Device
Description: Defined as mTICI 2b-3 flow in the target vessel post-treatment with the Q Catheter (first line therapy)
Time Frame: intra-procedural
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 38
Participants | 25

4. Secondary Outcome: Rate of Embolization to a New Neurovascular Territory (ENT)
Description: As measured by independent Angiographic Core Lab
Time Frame: intra-procedural
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Participants | 0

5. Secondary Outcome: Good Functional Outcome Measured by Modified Rankin Scale Score of 0-2
Description: The Modified Rankin Scale (mRS) measures neurological disability or dependence for stroke patients on a scale of 0 (no symptoms) to 6 (deceased).
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Participants | 25

6. Secondary Outcome: Mortality Rate
Description: Rate of all cause mortality
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Q Aspiration Catheter
Number analyzed (Participants) | 45
Participants | 7

ADVERSE EVENTS:
Time Frame: From procedure through subject 3 month follow up visit, serious adverse events were collected
Arm/Group | Q Aspiration Catheter
All-Cause Mortality (participants affected / at risk) | 7/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 6/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q Aspiration Catheter (N=45)
Hemorrhagic transformation (General disorders) | 6 (6)
Death of unknown cause (General disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 1 (1)
mechanical ventilation complications (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Q Aspiration Catheter (N=45)
procedural complication (Injury, poisoning and procedural complications) | 6 (6) — vasospasm, vessel dissection, and/or access site complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04089917/Prot_SAP_000.pdf